CLINICAL TRIAL: NCT00188357
Title: HIPP Learning to Live Better With Lupus: The Health Improvement and Prevention Program in Systemic Lupus Erythematosus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); The Arthritis Society, Canada (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 03-0605-A; 03-0084
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2007-02-14 (Estimated); Status verified 2005-09

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Educational Status

INTERVENTIONS:
Behavioral: Education

SUMMARY:
Several studies have shown that persons with systemic lupus erythematosus (SLE) have poor general health and a higher risk of heart attack and bone loss (osteoporosis) compared to the general population. Some of the risks associated with heart attacks and bone loss are modifiable (can be changed). For example, high blood pressure, high cholesterol, smoking, lack of exercise are risk factors associated with heart attacks that can be changed. Whereas, age and a family history of heart attacks are risk factors that can not be changed. Similarly, a diet low in calcium, smoking and lack of exercise are modifiable risk factors associated with osteoporosis; while, family history and age are not modifiable. The Health Improvement and Prevention Program (HIPP) in Systemic Lupus Erythematosus was developed to increase the general health in persons who have lupus and to help reduce the risk of heart attacks and bone loss. This intervention program gives comprehensive

information about lupus and provides tools on how to live better with lupus. The program includes visits with a nurse case manager who will work in close collaboration with the lupus team. She will work on an individual basis with each participant to develop a mutually agreed upon personalized care plan aimed at improving general health, coping skills and heart and bone health.

HIPP STUDY (Health Improvement And Prevention Program)

Dr Paul Fortin Principal Investigator

Primary and Secondary objectives:

* To improve health status, decrease cardiovascular risk and improve endothelial function in persons with SLE compared to usual care.
* To improve bone health behaviors and prevent decrease in bone mineral density.
* To improve adherence to treatments.
* To help persons with Lupus move toward wellness by increasing knowledge.
* To show that HIPP is cost effective and could become standard care.

Duration: 2 years

Enrollment 240 patients

Study Design:

* Randomized prospective study of HIPP compared to usual care, patients will be crossed over at Mth 12. Data collected for 24 mths.
* Demographic, health status, cost, SLE knowledge, coping, cardiovascular and osteoporosis information will be collected.
* All patients will undergo clinical evaluation to measure disease activity, BMD (every 2 years) and Flow mediated Doppler (every year)
* HIPP now patients will attend 4 knowledge sessions, covering SLE, coping with chronic disease, cardiovascular disease in Lupus, bone health in Lupus.
* HIPP now patients will be followed by nurse coordinator and receive an individualized risk assessment, telephone follow-up, smoking cessation counseling. For those found at risk stress reduction (Mindfulness Based Stress Reduction) and or bone health program will be provided. Hipp now patients will attend Cardiac Rehabilitation Program at TWH. All HIPP now pts will attend the Cardiac Rehabilitation program at the TWH.

Inclusion Criteria:

SLE according to ACR, >18 yr, Female, must read and write french or english

Exclusion Criteria:

MI, TIA, CVA, Other arterial occlusion, PVD, Osteoporosis as defined by BMD, Pregnant now, active cancer

For further information contact Study Coordinator Anne Cymet Tel # 13-2895 Pager 416-664-

DETAILED DESCRIPTION:
The survival rate in Systemic Lupus Erythematosus (SLE) exceeds 90% at 10 years but health status is severely impaired and comparable with that of advanced cardiac or respiratory diseases. Since these issues are often overlooked in clinical practice and because SLE affects primarily young women in their productive life, a specific intervention is needed to heighten health status and coping, and to reduce complications such as cardiovascular diseases (CVD) and osteoporosis.

Our primary goal is to demonstrate: 1- that a coordinated intervention, named the Health Improvement and Prevention Program (HIPP), will improve health status in SLE compared with usual care, and 2- that the same intervention will decrease significantly the number of cardiovascular risk factors and improve the flow-mediated dilatation (FMD - a non-invasive measure of endothelial health that we will use as a surrogate marker of CVD) in persons with SLE. Our secondary goals are to demonstrate that HIPP will: 1- improve bone health behaviors and prevent decrease in bone mineral density (BMD), 2- improve adherence to treatments, 3- help persons with lupus move towards wellness on the illness-wellness continuum by increasing their knowledge of lupus, and 4- be shown to be a cost-effective intervention that could become standard of care in SLE.

Our population will consist of consecutive patients with a diagnosis of SLE (revised 1997 ACR criteria) from the lupus clinics of the University of Toronto and McGill University. All those without cardiovascular disease or osteoporosis will be approached for this study. These two centres follow annually a total of close to 700 persons with SLE and offer standard HIPP services.

Our study design is a randomized prospective study of HIPP compared to usual care. As we believe that HIPP will be superior to usual care, we will crossover those in the usual care group to the HIPP group at 12 months. We will collect information for 24 months on all participants. The Health Improvement and Prevention Program is a multidisciplinary intervention that will be coordinated by a case manager nurse in close collaboration with the lupus treating team. After providing consent, each person will fill in demographic, health status, cost, SLE knowledge, coping, cardiovascular and osteoporosis risk questionnaires and will undergo a clinical evaluation to measure lupus disease activity and damage as well as a FMD and BMD. They will be randomized to HIPP or to usual care for 12 months after which the usual care group will be crossed over to HIPP. HIPP participants will be invited to attend a 4-week, 6 hour course that will cover the following four topics: 1) Knowledge of SLE, 2) Coping with a Chronic Disease, 3) Cardiovascular Disease in SLE and 4) Bone Health in SLE. Four to six weeks after entry into HIPP, there will be a second visit to the case manager during which an individualized program will be proposed to the patient. For all patients, this will include a standardized CVD prevention program. For those found to be at risk at baseline, it will also include a stress-reduction and/or a bone-health program. The case manager will follow HIPP participants individually by phone or in person according to their needs. Follow-up questionnaires on health status, cost and coping will be done by phone at 6 and 18 months; repeat clinical assessments for lupus activity and damage, questionnaires and FMD will be done at 12 and 24 months; and BMD will be repeated at 24 months.

Power and analyses. We will need to enroll 120 patients in our study to ensure 80% power to detect at least a 10% improvement in the SF-36 MCS and PCS and a 20% CVD risk reduction. Descriptive analyses, univariate and multivariate analyses will be carried out. For our primary goals, we will test whether HIPP is better than usual care in improving the SF-36 MCS, PCS and CVD risk profile. Our outcome will be change in the SF-36 MCS or PCS scores, FMD or CVD risk assessment, and our predictive variable will be HIPP. We will adjust for age, gender, and baseline SF-36 MCS and PCS, depression score, education, lupus activity and damage. Other secondary outcomes will be analysed using similar models. Cost will be calculated and cost-effectiveness analyses of HIPP will be performed.

Significance. A valid, cost-effective and comprehensive program to ameliorate the health and coping status and to prevent CVD and osteoporosis would have a high impact on the long-term health and quality of life of persons with SLE.

ELIGIBILITY:
Inclusion Criteria:

SLE acording to ACR Criteria > 18 years Female Able to read and write English or French -

Exclusion Criteria:

- History of Angina Myocardial infarction Cerebral Vascular Accident other arterial occlusions Peripheral Vascular disease Osteoporosis with documented fracture Pregnancy or intention of in next year Cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360
Dates: Start 2003-08

PRIMARY OUTCOMES:
Coordinated intervention will improve health status of patients with Lupus compared with usual care
Intervention will significantly decrease the number of cardiovascular risk factors and will improve flow mediated dilatation ( a non invasive measure of edothelial health

SECONDARY OUTCOMES:
Improve bone health behaviours and prevent decrease in bone mineral density
improve adherance to treatments
help persons with lupus move toward on the illness-wellness continuum by increasing their knowledge of Lupus
cost effective intervention that could become standard of care in lupus

CONTACTS AND LOCATIONS:
Overall Officials: Paul R Fortin, MD,FRCP,MPH, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network Toronto Western Division, Toronto, Ontario, Canada